CLINICAL TRIAL: NCT02006394
Title: Novel Dietary Interventions for Treating Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dorothy Sears, Associate Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB #110549
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Insulin Resistance; Obesity; Metabolic Syndrome
Keywords: Inflammation; Monocytes
MeSH Terms: conditions — Insulin Resistance; Obesity; Metabolic Syndrome; Inflammation | interventions — Fish Oils; Polyphenols; Corn Oil; Starch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Diet (Experimental): Reduced glycemic index bread products, fish oil capsules, and polyphenol capsules.
  Interventions: Dietary Supplement: Fish Oil; Dietary Supplement: Polyphenol Capsules; Other: Reduced glycemic index bread products
- Placebo Diet (Placebo Comparator): Market variety bread products, corn oil capsules, and corn starch capsules.
  Interventions: Dietary Supplement: Corn Oil Capsules; Dietary Supplement: Corn starch capsules; Other: Market variety bread products

INTERVENTIONS:
Dietary Supplement: Fish Oil — fish oil capsules
  Arms: Active Diet
Dietary Supplement: Polyphenol Capsules — delphinidin polyphenol capsules
  Arms: Active Diet
Dietary Supplement: Corn Oil Capsules — Corn Oil Capsules
  Arms: Placebo Diet
Dietary Supplement: Corn starch capsules — Maltodextrin capsules
  Arms: Placebo Diet
Other: Reduced glycemic index bread products — Made by Zone Labs
  Arms: Active Diet
Other: Market variety bread products — placebo bread products
  Arms: Placebo Diet

SUMMARY:
Clinical and rodent studies have demonstrated the impact of specific dietary factors in modulating inflammation-related diseases including insulin resistance, type 2 diabetes, and cardiovascular disease. Such dietary factors include polyunsaturated fats, polyphenols, and glycemic index. The investigators know from previous studies in the literature that reducing the glycemic index and increasing the omega-3 fat and polyphenol content of the diet results in improved metabolic indices and reduced inflammation. These improvements can be observed even within the context of persistent obesity. The investigators will implement a reduced-calorie, multi-pronged dietary approach for improving insulin sensitivity and reducing inflammation in obese subjects with the metabolic syndrome. The active diet will include reduced glycemic index foods together with omega-3 fats and polyphenol supplements. The primary hypothesis is that the dietary combination of reduced glycemic index foods, omega-3 fats and polyphenols will work to reduce insulin resistance and inflammation more efficiently than a placebo-controlled, calorie- and macronutrient-matched diet in obese subjects with the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI): 30.0-40.9 kg/m^2
* Metabolic Syndrome

Exclusion Criteria:

* Diabetes
* Inflammatory diseases
* Eating disorders
* Pregnancy
* Known kidney, coronary, gastrointestinal or peripheral artery disease
* Smoking
* Recent fish oil (>500mg eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA)/day) or polyphenol supplement use
* Recent weight change
* Strenuous exercise
* Fish/food allergies
* Current diabetic, lipid-lowering (fibrates, statins), anti-inflammatory, immune-suppressant, and/or anti-inflammatory hypertension medication use

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in insulin resistance | Baseline, 6 weeks, and 12 weeks
  Fasting plasma insulin, Homeostasis Model of Assessment - Insulin Resistance (HOMA-IR)

SECONDARY OUTCOMES:
Change in inflammation biomarkers | Baseline, 6 weeks, 12 weeks
  Fasting plasma cytokines and C-reactive protein (CRP), monocyte expression of inflammatory genes

OTHER OUTCOMES:
Change in adipokines | Baseline, 6 weeks, 12 weeks
  Fasting plasma adiponectin and leptin

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Sears, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States